CLINICAL TRIAL: NCT04301219
Title: Knowledge and Practices of Adverse Drug Reaction Reporting Among Healthcare Professionals in Low and Middle-income Countries: a Cross-sectional Survey.
Brief Title: Knowledge and Practices of ADR Reporting in LMICs
Status: Completed | Type: Observational
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GTZ-PV-001
Record Dates: First submitted 2019-11-26; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Adverse Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The reported literature suggests that knowledge about pharmacovigilance is on a lower side and ADR reporting is not common in developing countries. This survey may help us to identify the common gaps in knowledge and practices about pharmacovigilance so that we can devise the strategy on the basis of outcome.

DETAILED DESCRIPTION:
Safety evaluation of a product in a market is like a moving ball which need re-evaluation as the data gather in its life cycle.(1) As per the definition of International society of harmonization and World Health Organization, adverse reaction is Adverse drug reaction (ADR) is defined as "A response to a drug which is noxious and unintended and which occurs at doses normally used in man for prophylaxis, diagnosis, or therapy of disease or for modification of physiological function." (2) Adverse reaction and adverse event are interchangeable use in pharmacovigilance sector by knowing the difference is that ADR term used when drug is causing the effect (1). The frequency of ADR is getting higher due to the increasing prevalence of chronic disease with the growing trend of combination drugs (3). The non-profitable organization of pharmacovigilance is playing tremendous role in disseminating the awareness of proper usage of drug globally.(3) According to Uppsala database statistics, approximately 3 million reports were listed as suspected ADRs. (4) Nearly 6.7% of hospitalizations were due to serious ADRs (5)

ELIGIBILITY:
Inclusion Criteria:

- Participants who would like to voluntarily fill the survey form

Exclusion Criteria:

* Students
* Other than Health care professionals (including but not limited to Physicians, Doctors, Nurses and/or pharmacist)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A self-administered questionnaire was distributed to 1500 HCPs in 11 countries (Afghanistan, Cambodia, Kazakhstan, Kenya, Laos, Myanmar, Nigeria, Pakistan, Philippines, Sri Lanka, and Sudan). The participants were approached at various scientific events and academic interactions during the period and were requested to participate in the survey on a voluntary basis.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Country-wise Analysis on knowledge of HCPs | 2 years
  Number of HCPs had knowledge about AR in their own country
Country-wise Analysis on practices of HCPs | 2 years
  Number of HCPs practicing AR reporting in their own country

CONTACTS AND LOCATIONS:
Overall Officials: Mahwish Raza, Pharm-D, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University, Karachi, Sindh, Pakistan